CLINICAL TRIAL: NCT01671618
Title: A Prospective Study on Point-of-Care Focused Cardiac Ultrasound in Assessing for Thoracic Aortic Dimensions, Dilation, and Aneurysm in Correlation With CT Angiogram in Suspected Cases of Pathology
Brief Title: Point-of-Care Focused Cardiac Ultrasound in Assessing the Thoracic Aorta
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1202009791
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Aortic Aneurysm, Thoracic; Aortic Dissection
Keywords: Aortic dissection; Aortic dilation; Aortic Aneurysm; ultrasound; point-of-care; echocardiography
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Aortic Dissection; Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this prospective study is to compare point-of-care focused cardiac ultrasound (FOCUS) to thoracic computed tomographic angiography (CTA) in the measurement of ascending aortic dimensions. We hypothesize that FOCUS will demonstrate good agreement with CTA in the measurement of ascending aortic dimensions and accurately detect dilation and aneurysmal disease.

DETAILED DESCRIPTION:
Nonspecific chest pain is frequently encountered in the emergency department. Accounting for over 13,000 deaths annually, aortic aneurysmal disease is a potential cause of chest pain.There are multiple diagnostic imaging modalities in practice to interrogate the thoracic aorta, with the most common being computed tomographic angiography (CTA), trans-thoracic echocardiography (TTE) and trans-esophageal echocardiography (TEE), each with its own advantages and limitations. In the ED setting, point-of-care (POC) focused cardiac ultrasound (FOCUS) is increasingly being used as an adjunct to the emergency physician's (EP) workup of undifferentiated chest pain. Based on prior retrospective data FOCUS and CTA appear to have good agreement. This studies aims to confirm these findings through prospective evaluation

Specific Aims

Aim 1: To prospectively compare Point of Care (POC) Focused Cardiac Ultrasound (FOCUS) to thoracic computed tomographic angiography (CTA) in the measurement of ascending aortic dimensions.

Maximal diameter measurements of the ascending thoracic aorta by FOCUS will be compared to CTA. Bland Altman plots with 95% limits of agreement will be used to determine clinical and statistical significance.

Hypothesis: 95% limits of agreement between FOCUS and CTA will be within +/- 5 mm.

Aim 2: To determine the diagnostic accuracy of Point-of-Care Focused Cardiac Ultrasound for the detection of thoracic aortic dilation and aneurysm with computed tomographic angiography as the reference standard

Sensitivity, Specificity and Accuracy of FOCUS will be computed with CTA as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years and older presenting to the ED for whom a thoracic CTA has been ordered.

Exclusion Criteria:

* Refusal of verbal consent for ultrasound.
* Inability to obtain informed written consent for data collection from either the patient or the patients decision-making surrogate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older presenting to an urban, academic, and level I emergency department with estimated volume of approximately 90,000 patients per year.
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Maximal diameter measurements of the proximal ascending aorta by CTA and FOCUS | during emergency department visit (estimated average 3-6 hours)
  Maximal diameter measurements of the ascending thoracic aorta by FOCUS will be compared to CTA. Bland Altman plots with 95% limits of agreement will be used to determine clinical and statistical significance.

SECONDARY OUTCOMES:
Time to Emergency Department Disposition | estimated time frame 3-6 hours
  Time until an admission or discharge order is placed within the electronic medical record
Number and percent probabilities of differential diagnosis | (estimated time frame 0 -3 hours)
  Number and percent probabilities of differential diagnosis will be obtained before and after ultrasound to calculate the informational content provided by the ultrasound and perform additional uncertainty analyses
Time to diagnostic imaging | estimated time frame 0-6 hours
  Time when diagnostic imaging is performed

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Taylor, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States